CLINICAL TRIAL: NCT05450094
Title: Patient-Centered Enhancements to Reduce Unmet Mental Health Need of African-American Children
Brief Title: Reducing Unmet Mental Health Need of African-American Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202200678; AD-2021C1-22495 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): The comparator arm enhances school-based mental health (SBMH) with universal screening and trains voluntary school teams to use the school-wide data to plan and make intervention referrals using an evidence-based in-service training and coaching model called Team-Initiated Problem Solving (TIPS).
  Interventions: Behavioral: Screening Only
- Enhanced (Experimental): The enhanced arm involves the enhancements to school-based mental health (SBMH) of the comparator arm with the addition of 3 additional empirically-based implementation supports, including training, coaching, and data-based feedback. Enhancement aim to increase school teams' awareness and understanding of students' mental health well-being and need for intervention.
  Interventions: Behavioral: Enhanced Screening

INTERVENTIONS:
Behavioral: Screening Only — The Screening Only intervention integrates enhancements to school-based mental health (SBMH). Each school's typical SBMH service delivery system will be enhanced with biweekly meetings of voluntary school teams (comprised of administrators, school counselors, general and special education teachers, and other school-employed mental health professionals) to 1) follow standardized evidence-based intervention decision making process to identify students with mental health risk, plan and/or refer for an evidence-based intervention, monitor intervention progress, and adjust intervention plans as needed; 2) administer teacher-rated and student self-report universal screening twice annually; 3) review screening and related school records data to identify students with mental health risk; and 4) review screening, referral, and receipt data to monitor progress of entire SBMH service delivery system.
  Arms: Comparator
Behavioral: Enhanced Screening — The Enhanced Screening intervention involves the enhancements to school-based mental health (SBMH) of the Screening Only intervention with the addition of 3 empirically-based implementation supports, including training, coaching, and data-based feedback. Enhancement aim to increase school teams' awareness and understanding of students' mental health well-being and need for intervention. enhancements.
  Arms: Enhanced

SUMMARY:
The purpose of this study is to compare two versions of school-based mental health screening to improve the receipt of mental health services among elementary school students.

DETAILED DESCRIPTION:
School-based mental health (SBMH) is a critical pathway for accessing mental health services for African American/Black (AAB) youth who experience the greatest gap in unmet mental health need in comparison to their White, non-Hispanic peers, but are twice as likely to access mental health services in schools as outpatient or specialty clinics. Unfortunately, AAB children's access to SBMH is dependent on school intervention team decision making, which often involves consideration of factors other than student need. School personnel on intervention teams disproportionately attribute AAB youth's behavior problems as disciplinary issues rather than mental health needs, reducing the likelihood AAB students receive SBMH services. Consistent with the empirical literature, patient families and stakeholders recommend universal mental health screening to better identify AAB children with mental health needs and enhancements to address implicit social cognitions that impact decision-making processes and poor mental health literacy of school personnel making intervention referral decisions. Thus, we will evaluate the comparative effectiveness of the SBMH delivery system enhanced with screening to a package of enhancements implemented with screening in SBMH to increase the likelihood AAB students receive the services they critically need. The enhancements include implementation supports, including training, coaching, and data-based feedback. We will test both whether and how (i.e., mediational analyses of causal pathway including knowledge, attitudinal, and behavioral observation of unintentional bias and mental health literacy) these enhancements impact student-level intervention and disciplinary referral outcomes. In a mixed method process evaluation and comparative analysis, we will also examine school-level contextual factors (i.e., team member tenure, pre-intervention discipline rates, racial/ethnic and socioeconomic composition of student body, and perceptions of intervention impact and acceptability) and implementation outcomes (i.e., fidelity, dosage/exposure, and reach).

ELIGIBILITY:
Inclusion Criteria:

* Students at study school
* School intervention teams at study school

Exclusion Criteria:

* Students who are wards of the state or any other institution, agency, or entity

Ages: 5 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19106 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in student referral to a mental health intervention as measured by the number of students referred to mental health interventions each quarter | From first day of school in year 1 to last day of school in year 2
  Intervention referrals refer a student to a mental health intervention to address an identified mental health need. The number of students referred to a mental health intervention will be counted. The minimum score is 0 and there is no maximum score.

SECONDARY OUTCOMES:
Mean change from baseline in student disciplinary encounters as measured by the number of Office Discipline Referrals each quarter | From first day of school in year 1 to last day of school in year 2
  Office Discipline Referrals are official school records recorded for each school behavioral infraction warranting referral to the school office. Office Discipline referrals for aggressive behavior (i.e. bullying, fighting, making threats) will be counted. The minimum score is 0 and there is no maximum score.

CONTACTS AND LOCATIONS:
Overall Officials: Joni Splett, Ph.D, Principal Investigator — University of Florida
Locations (1):
- Name withheld to protect anonymity of study site, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Splett JW, Gage NA, Chaparro EA, Lyon AR, Sonsteng-Person MA, Alfonso ZZ, Halliday CA. Differential item functioning of teacher-rated universal mental health screening in elementary schools. Sch Psychol. 2025 Sep 29. doi: 10.1037/spq0000712. Online ahead of print. PMID 41021530